CLINICAL TRIAL: NCT04534608
Title: Prevalence of Infection and Seroconversion and the Clinical Course of the Novel Coronavirus SARS-CoV-2 Infection in Children Between 0 to 18 Years of Age in Hamburg and Surroundings
Brief Title: COVID-19 Child Health Investigation of Latent Disease in Hamburg
Acronym: C19CHILD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Altona Children's Hospital (Other); Wilhelmstift Children´s Hospital (Unknown); Helios Mariahilf Klinik Hamburg (Unknown); Asklepios Klinik Nord - Heidberg (Unknown)
Responsible Party: Principal Investigator, Ania C. Muntau, Medical Director, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: PV7336
Record Dates: First submitted 2020-08-31; First posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: SARS-CoV-2; Covid19
Keywords: pediatric; children; observational; antibody; PCR; immunology; metabolomics; household
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Asymptomatic children w/out an underlying condition
- Asymptomatic children with underlying condition(s)
- Children with COVID-19 symptoms w/out an underlying condition
- Children with COVID-19 symptoms with underlying condition(s)

SUMMARY:
The study measures infection rates and the presence of antibodies for SARS-CoV-2 (COVID-19) among in- and outpatients of all pediatric hospitals, as well as volunteers aged 0 to 18 years in Hamburg, Germany. Participants with a positive nasopharyngeal swab PCR or a positive antibody test enter the Follow-up phase of 6 months. The follow up includes a PCR and antibody testing of all household contacts at 0, 3 and 6 months, as well as laboratory testing of children to identify immunological, metabolic and genetic risk factors for infection and clinical outcome.

DETAILED DESCRIPTION:
The study is divided into a Screening phase and a Follow-up phase. In the Screening phase, an obligatory polymerase chain reaction (PCR) in the nasopharyngeal swab and an optional serum antibody testing are carried out for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). An obligatory standardized questionnaire is used to evaluate symptoms and contacts, medical history and underlying conditions and the psychological effects of the Coronavirus disease 2019 (COVID-19) pandemic, as well as its effects on individual access to medical care. Children with a positive nasopharyngeal swab or antibody test, as well as their household contacts aged 0 to 18 years enter the Follow-up phase. During the Follow-up phase, blood and urine samples are taken from children for immunological analysis, HLA typing and untargeted metabolomics, enabling a broad analysis of the adaptive and innate immune response to SARS-CoV-2, as well as metabolic and genetic risk factors for infection and disease compared to age and sex-matched healthy controls. Furthermore, a repeated swab and antibody testing at 0, 3 and 6 months for children and adult household contacts is carried out to analyse household transmission of SARS-CoV-2 in children and adults and the persistence of antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Children or Teenagers aged 0-18 years
* Patient in one of the participating centers or volunteer in the central C19.CHILD Study Clinic
* Informed consent from parents or guardians.
* Informed consent from children >7 years (unless not capable)

Exclusion Criteria:

* Prematurity <37 weeks of gestation
* Informed consent of parents and guardians not possible in spoken word or otherwise
* Informed consent not given

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 1. In- and outpatients aged 0 to 18 years of all pediatric hospitals in Hamburg, Germany
  2. Healthy children aged 0 to 18 years as volunteers
  3. Participants of other studies or their children (Prenatal Investigation of Children's Health - PRINCE Study, Hamburg City Health Study)
  4. Children, who are household contacts of SARS-CoV-2 positive study participants will directly enter the Follow-up phase
  Healthy Control Group:
  A group of children tested negative for SARS-CoV-2 by PCR and antibody testing will be included as control group for the immunologic, metabolic and genetic follow up. This group is recruited from participants in group 2 and 3 (above).
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Acute infection by SARS-CoV-2 | 6 weeks
  Detection of SARS-CoV-2 by PCR in the nasopharyngeal swab

SECONDARY OUTCOMES:
Seroconversion for SARS-CoV-2 | 6 months
  Detection of antibodies against SARS-CoV-2 in serum
Immune phenotyping | 6 months
  Analysis of the innate and adaptive immune system by flow cytometry
HLA Typing | 6 months
  HLA typing by sequencing to identify protective- and risk constellations
Matabolomics | 6 months
  Untargeted metabolomics in urine and plasma

CONTACTS AND LOCATIONS:
Overall Officials: Ania C Muntau, Professor, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Soeren W Gersting, Professor, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Thomas Mir, Professor, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Universitätsklinikum Hamburg-Eppendorf, Department of Pediatrics Homepage — https://www.uke.de/kliniken-institute/kliniken/kinder-und-jugendmedizin/index.html